CLINICAL TRIAL: NCT04284124
Title: Erector Spinae Block Versus PECS Block Type II for Breast Surgeries: a Randomized Controlled Trial
Brief Title: Erector Spinae Block Versus PECS Block Type II for Breast Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Bakir, Assistant Professor of Anesthesia, Intensive care and Pain relief, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AP2001-50504
Record Dates: First submitted 2020-02-18; First posted 2020-02-25 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae block (Active Comparator): Done unilaterally with the patient in the prone position about 20 min before induction of general anesthesia. Skin is prepared by 10% povidone iodine. An ultrasound machine with a large bandwidth, multifrequency convex probe (1-8 MHz) will be used for block performance. A 22G, 50-mm, at the T4 level of the spine using an in-plane approach. Probe is placed 2-3 cm laterally to the spine using a sagittal approach. Once the erector spinae muscle and the transverse processes is identified, the needle will be inserted deep into the muscle. The needle will be directed from a cranial to a caudal direction. Following confirmation of the correct position of the needle tip with administration of 0.5-1 ml of local anesthetic, 20 ml of 0.25% bupivacaine will be administered for block performance. Distribution of local anesthetic will be observed in both cranial and caudal directions.
  Interventions: Other: Erector Spinae block
- PECS type II block (Active Comparator): Done unilaterally, patient is put in the supine position with ipsilateral arm abducted and externally rotated with elbow flexed 90 degrees. High frequency probe is put in the ipsilateral clavipectoral triangle between the clavicle medially and above and the shoulder joint laterally. The pectoralis major and minor and the plane between them are identified guided by pulsating thoracoacromial artery or its pectoral branch. Needle is advanced in plane targeting the space where the artery is located, 2ml of normal saline is injected to confirm the location. Then, 10 ml of bupivacaine 0.25% is injected. Probe is moved laterally and caudally towards the anterior axillary fold parallel to the deltopectoral groove till the serratus muscle slips appear underneath the pec minor attached to the underlying ribs. Targeting the plane between pec minor and serratus at the level of the third rib, 2 ml of normal saline is injected for confirmation of the needle tip then 20 ml of bupivacaine 0.25%.
  Interventions: Other: Erector Spinae block

INTERVENTIONS:
Other: Erector Spinae block — Patient in the prone position 20 min before induction of general anesthesia. Skin is sterilized by 10% povidone iodine. An US multifrequency convex probe (1-8 MHz) will be used for block. A 22G, 50-mm in length needle will be used and block will be performed at the T4 level of the spine using in-plane approach where a convex probe is placed 2-3 cm lateral to the spine using sagittal approach. Erector spinae muscle and the transverse processes are located and the needle will be inserted deep into the muscle. The needle is directed craniotomy-caudally. Correct position of the needle tip is confirmed with administration of 0.5-1 ml of local anesthetic to monitor spread then 20 ml of 0.25% bupivacaine will be administered for block performance. Distribution of local anesthetic is monitored in both cranial and caudal directions

SUMMARY:
The purpose of this randomized, controlled prospective study is to compare the analgesic effect of US-guided ESP block versus PECs block in patients undergoing breast surgery for breast cancer in the National Cancer Institute, Cairo University. We aim to evaluate the postoperative pain intensity and opioid consumption within 24 hours

DETAILED DESCRIPTION:
This prospective, randomized controlled trial will include 30 adult female patients below 65 years of age scheduled for surgery for breast cancer. Inclusion criteria will include also American Society of Anesthesiologists (ASA) physical status I-II and unilateral surgery. Exclusion criteria will include obesity defined as body mass index > 35 kg/m2), known allergy to the study drugs, coagulopathy, skin infection at the site of needle puncture, and recent use of opioid drugs.

Patients will be assessed the day before surgery in a preoperative visit for evaluation of their medical status and laboratory investigations. They will be informed about the technique of the blocks and written informed consents will be obtained. All patients will be informed how to report pain on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain). In the pre-anesthetic room, midazolam 0.02 mg/kg IV will be given to the patients for sedation after fixation of a 20 G cannula as an IV line. Randomization will be done using consecutively numbered opaque sealed envelopes. Patients will be randomized into two groups according to the type of analgesia. The first group will receive single-shot ESP block (ESP group) and the other group will receive PECs II block (PECs group).

ESP technique:

ESP block will be performed in following standardized monitoring, including noninvasive blood pressure, electrocardiogram, and pulse oximetry. It will be done unilaterally with the patient in the prone position about 20 min before induction of general anesthesia. Skin is prepared by 10% povidone iodine. The US probe will be covered with a sterile cover. All blocks will be by the same anesthesiologists who are experienced in US-guided nerve blocks. An ultrasound machine with a large bandwidth, multifrequency convex probe (1-8 MHz) will be used for block performance. A 22G, 50-mm, insulated facet type needle will be used during all blocks. The blocks will be performed at the T4 level of the spine using an in-plane approach. A convex probe will be placed 2-3 cm laterally to the spine using a sagittal approach. Once the erector spinae muscle and the transverse processes is identified, the needle will be inserted deep into the muscle. The needle will be directed from a cranial to a caudal direction. Following confirmation of the correct position of the needle tip with administration of 0.5-1 ml of local anesthetic, 20 ml of 0.25% bupivacaine will be administered for block performance. Distribution of local anesthetic will be observed in both cranial and caudal directions.

PECs II block Technique:

The block will be done unilaterally about 20 min before induction of general anesthesia. Under standardized monitoring, the patient is put in the supine position with the ipsilateral arm abducted and externally rotated and the elbow flexed 90 degrees. The skin over the ipsilateral clavicle and small area below it is done by betadine. The high frequency probe is put in the ipsilateral clavipectoral triangle between the clavicle medially and above and the shoulder joint laterally. The pectoralis major and minor and the plane between them are identified. The probe is tilted caudally to identify the pulsating thoracoacromial artery or its pectoral branch. The skin at the point of entry is infiltrated by xylocaine 1% then the needle is advanced in an in plane technique targeting the space in which the artery is located. Two cm of normal saline is injected to confirm the location and produce dissection. Then, 10 ml of bupivacaine 0.25% with epinephrine 2.5 µg/ml is injected. Propofol is given in 20 mg boluses followed by normal saline flush to produce more sedation just before injecting the bupivacaine because dissection is painful. Then the probe is moved laterally and caudally towards the anterior axillary fold parallel to the deltopectoral groove till the serratus muscle slips appear underneath the pec minor attached to the underlying ribs. The 3rd and 4th ribs and the pleura are identified. After infiltration of the skin with xylocaine 1% the needle is advanced in plane targeting the plane between pec minor and serratus at the level of the third rib. Two ml of normal saline is injected for confirmation of the needle tip then 20 ml of bupivacaine 0.25% with epinephrine 2.5 µg /ml is injected. A pinprick test is done after 15 minutes to assess sensory block compared to the unblocked contralateral side. A block is considered unsuccessful and the patient is excluded from the study if the site of surgical incision is not blocked after 20 min of LA injection.

General anesthesia Standard anesthesia monitoring will be applied, and induction of general anesthesia will be carried out by using fentanyl (1µg/kg) IV, propofol (2 mg/kg) IV and cisatracurium (0.15mg/kg) IV. Paracetamol 1 gm/100 ml IV infusion and ketolac 30 mg IV slowly is given before surgical incision. Paracetamol 1 gm/100 ml IV infusion is given every 8 hours and ketolac 30 mg every 12 hours. Anesthesia will be maintained by sevoflurane 2% in O2 and supplemental doses of cisatracurium (0.03 mg/kg) IV as indicated by peripheral nerve stimulator by appearance of the second twitch of the train of four (TOF). Additional bolus doses of fentanyl 0.5 µg /kg will be given if the mean arterial blood pressure and/or heart rate rise above 20% of baseline. The patients will receive fluids in order to replace their fluid deficit, maintenance and losses, and will be mechanically ventilated at appropriate setting that keep end-tidal CO2 at 30-35 mmHg. Hypotension will be treated with 0.9% normal saline, 6% hetastarch in saline and/or 5mg ephedrine in incremental doses in order to maintain mean blood pressure above 70 mmHg. Recovery will be carried out after closure of surgical wound by turning off sevoflurane vaporizer and reversal will be given after TOF ratio becomes 0.7 and fully awake extubation will be done and then the patient will be transferred to post anesthesia care unit (PACU)

In the PACU, VAS is assessed by a nurse blinded to the intervention done. It will be assessed immediately postoperative, and then 1, 2, 6, 12, and 24 hours post-extubation. Patients will be given 2 mg morphine slowly IV when VAS > 3, repeated 2 times if required (total 3 boluses) to keep VAS ≤ 3, at least 10 minutes between each bolus, then 1 mg morphine is given slowly IV if required, at least 15 minutes between each bolus. Nausea and/or vomiting are treated by metoclopramide 10 mg/8 hours slowly IV. Incidences of nausea and vomiting, and total morphine consumption during the 24-h postoperative period were recorded.

The primary outcome measure of the study will be total morphine consumption during the first 24 postoperative hours. The secondary outcome measures will be duration of analgesia, postoperative pain scores up to 24 hours postoperative, and occurrence of postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Adult patients (>18 years old)
* Female sex
* Scheduled for breast surgeries at NCI, CU

Exclusion Criteria:

* Patient's refusal of the study procedures
* Allergy to drugs used in the study
* Patients with chronic pain and chronic use of opioids
* Patients with coagulopathies (INR > 1.6 or platelets count < 50,000 cc3)
* Hemodynamically unstable patients (e.g. BP < 90/60)
* Patients with local or systemic infections concerning intervention sites and septic patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is performed on female patients undergoing breast surgeries after diagnosis with breast cancer
Enrollment: 60 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption for 24 hours post operatively | 24 hours
  The primary outcome measure of the study will be total morphine consumption during the first 24 postoperative hours.

SECONDARY OUTCOMES:
duration of analgesia | 24 hours
  duration of analgesia post operatively
post operative pain scores using numerical rating scale | 24 hours
  post operative pain scores using numerical rating scale (NRS) for 24 hours with 0 to no pain and 10 to most severe pain
post operative nausea and vomiting using nausea score | 24 hours
  post operative nausea and vomiting for 24 hours using nausea score with 0 for no nausea, 1 for mild nausea, 2 for moderate nausea, 3 for severe nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Bakir, M.D, Principal Investigator — NCI Egypt
Locations (1):
- NCI Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided